CLINICAL TRIAL: NCT03428724
Title: A Randomized Clinical Trial Comparing Standard and Invidualized Bowel Preparation for Colonoscopy
Brief Title: Individualized Bowel Preparation for Colonoscopy
Acronym: PREP2TARGET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, dr. Theodor Alexandru Voiosu, MD, PhD, Clinical Hospital Colentina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COL-GASTRO-6
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Colon Disease
MeSH Terms: conditions — Colonic Diseases | interventions — Reference Standards

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard group (Active Comparator): standard polyethylene glycol preparation for colonoscopy
  Interventions: Drug: Standard Preparation
- individualized group (Experimental): either a low or a high volume bowel preparation according to patient characteristics
  Interventions: Drug: Individualized Preparation

INTERVENTIONS:
Drug: Standard Preparation — standard PEG-based bowel preparation for colonoscopy (either split dose 4L polyethylene glycol or split 2L PEG + ascorbic acid)
  Arms: standard group
Drug: Individualized Preparation — individualized bowel preparation for colonoscopy (either split dose 4L PEG or split 2L PEG + ascorbic acid) based o patient characteristics (history of failed bowel preparation; use of laxative drugs, increased BMI, age>65, neurologic comorbidities)
  Arms: individualized group

SUMMARY:
A randomized control trial comparing a standard bowel preparation for colonoscopy with an individualized bowel preparation strategy based on patient characteristics

ELIGIBILITY:
Inclusion Criteria:

* elective out-patient diagnostic or therapeutic colonoscopy

Exclusion Criteria:

* pregnant women; refusal to participate; significant comorbidities (ASA score 3 or above); suspicion of bowel perforation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
bowel preparation quality | 1-2 hours after completing bowel preparation
  Boston bowel preparation score (BBPS)

SECONDARY OUTCOMES:
patient comfort during bowel preparation | 1-2 hours after completing bowel preparation
  0-10 patient comfort score using a standard visual-analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Theodor Voiosu, Principal Investigator — Clinical Hospital Colentina
Locations (2):
- Romania (2):
  - Colentina Clinical Hospital, Bucharest
  - Carol Davila Emergency Military Hospital, Bucharest